CLINICAL TRIAL: NCT01351454
Title: Behavioral Depression Treatment for African American HIV-infected Substance Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-0341; R01DA026424 (NIH); R01DA022974 (NIH)
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Depression; Substance Use
Keywords: Depression; Substance Use; HIV Medication Adherence; Behavioral Activation
MeSH Terms: conditions — Depression; Substance-Related Disorders | interventions — Person-Centered Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACT HEALTHY (Active Comparator): ACT HEALTHY is based on the empirically validated Behavioral Activation Treatment for Depression (BAT-D; Lejuez, Hopko, & Hopko, 2001) and Life Steps, an HIV medication adherence intervention (Safren, Otto, & Worth, 1999). ACT HEALTHY is based on the belief that the best way to improve mood, remain sober, increase medication adherence, and make long-term life changes is by changing and increasing one's activity level. Treatment includes 16 individual sessions over a 12-week period.
  Interventions: Behavioral: ACT HEALTHY
- Nondirective Therapy (NDT) (Placebo Comparator): In NDT, the therapist will create an accepting, nonjudgmental, empathic environment to continuously direct client attention to primary feelings, and to facilitate accepting of affective experience using supportive statements, reflective listening, and empathic communications. In addition, medication adherence is addressed with the Life Steps HIV medication adherence intervention (Safren, Otto, & Worth, 1999). Treatment includes 16 individual sessions over a 12-week period.
  Interventions: Behavioral: Nondirective Therapy (NDT)

INTERVENTIONS:
Behavioral: ACT HEALTHY — ACT HEALTHY is based on the empirically validated Behavioral Activation Treatment for Depression (BAT-D; Lejuez, Hopko, & Hopko, 2001) and Life Steps, an HIV medication adherence intervention (Safren, Otto, & Worth, 1999). ACT HEALTHY is based on the belief that the best way to improve mood, remain sober, increase medication adherence, and make long-term life changes is by changing and increasing one's activity level. Treatment includes 16 individual sessions over a 12-week period.
  Other Names: LETS ACT; Behavioral Activation; Life Steps
  Arms: ACT HEALTHY
Behavioral: Nondirective Therapy (NDT) — In NDT, the therapist will create an accepting, nonjudgmental, empathic environment to continuously direct client attention to primary feelings, and to facilitate accepting of affective experience using supportive statements, reflective listening, and empathic communications. In addition, medication adherence is addressed with the Life Steps HIV medication adherence intervention (Safren, Otto, & Worth, 1999). Treatment includes 16 individual sessions over a 12-week period.
  Other Names: Supportive Counseling; Life Steps
  Arms: Nondirective Therapy (NDT)

SUMMARY:
The objective of the current study is to test a novel, behavioral approach to treat depressive symptoms and improve HIV medication adherence and subsequent physical health outcomes among African American HIV-infected substance users residing in inner-city Washington, DC. This treatment will serve as a compliment to standard residential and follow-up outpatient substance use treatment, with the goal of reducing depressive symptoms and improving HIV medication adherence, physical health, and substance use outcomes.

DETAILED DESCRIPTION:
Approximately 37-50% of HIV positive individuals suffer from depression, which is associated with substance use, poor adherence to HIV medication, an increase in HIV risk behaviors, and subsequent poor health outcomes (e.g., Asch et al., 2003; Bing et al., 2001; Dew et al., 1997; Johnson, Rabkin, Lipsitz, Williams, & Remien, 1999). Additionally, depressed HIV positive substance users are at an even greater risk for poor medication adherence than non-substance users (Cook, Grey, & Burke-Miller, 2004). Notably, evidence indicates that HIV positive patients who receive treatment for depression exhibit significant improvements in HIV medication adherence and a reduction in risk behaviors that are directly relevant to their health and well being such as risky sexual behavior (e.g., Cook et al., 2006). Despite this link, few interventions targeting depression have been developed to meet the specific needs of HIV-infected substance users. This is especially evident for low income African American HIV positive substance users who often do not receive adequate treatment for any of these conditions due to poverty, lack of access to specialized treatment, low motivation, cognitive impairments, and a lack of coordination between medical, mental health, and substance abuse treatment providers (Calsyn et al., 2004). Thus, the objective of the present proposal is to test a novel, behavioral approach to treat depressive symptoms and improve HIV medication adherence and subsequent physical health outcomes among African American HIV infected substance users residing in inner-city Washington, DC. This treatment combines (1) LET'S ACT, a behavioral activation based treatment for depressed substance users (Daughters, Braun, Sargeant, Hopko, Blanco, & Lejuez, 2008), with (2) Life Steps, an HIV medication adherence intervention (Safren, Otto, & Worth, 1999). The purpose of this combined treatment will be to compliment standard residential and follow-up outpatient substance use treatment to specifically treat depressive symptoms with the additional goal of improving HIV medication adherence, substance use, and physical health outcomes. Participants will be randomly assigned to either treatment as usual (TAU) plus ACT HEALTHY or TAU plus Nondirective Therapy to test the efficacy of ACT HEALTHY. Treatment as usual for both groups consists of standard residential and outpatient substance abuse treatment. Based on the outcome of this preliminary trial, the ACT HEALTHY protocol will be further refined and readied for larger-scale clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years of age
* HIV positive

Exclusion Criteria:

* psychosis
* the inability to give informed, voluntary, written consent to participate
* reading ability [below 3rd grade level on the WRAT]

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI-II; Beck et al., 1996) | BDI-II will be evaluated from baseline to a 12-month follow up period
  The Beck Depression Inventory is a 21-item self-report measure of depressive symptoms.
MEMS | MEMS is assessed from residential discharge to 12-month follow up period
  The MEMS cap (AARDEX) is an electronic pill bottle designed to record HIV medication adherence.
Urinalysis | Urinalysis is assessed from residential discharged to a 12-month follow up period
  Urinalysis is a biological measure of substance use.
Time Line Follow Back (TLFB) | TLFB will be assessed from baseline to a 12-month follow up period
  The Time Line Follow Back is a self-report measure of drug and alcohol use.
Adherence to Anti-Retroviral Medications Questionnaire (ACTG; Chesney, Morin, & Sherr, 2000) | ACTG will be assessed from baseline to 12-month follow up period
  The ACTG is self-report measure of HIV medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey B. Daughters, Ph.D, Principal Investigator — University of Maryland, College Park
Locations (2):
- United States (2):
  - Salvation Army Harbor Light Treatment Center, Washington D.C., District of Columbia
  - University of Maryland, College Park, Maryland

REFERENCES:
- [Background] Daughters SB, Magidson JF, Schuster RM, Safren SA. ACT HEALTHY: A Combined Cognitive-Behavioral Depression and Medication Adherence Treatment for HIV-Infected Substance Users. Cogn Behav Pract. 2010 Aug 1;17(3):309-321. doi: 10.1016/j.cbpra.2009.12.003. PMID 21709737
- [Derived] Belus JM, Tralka H, Satinsky EN, Seitz-Brown CJ, Daughters SB, Magidson JF. Substance Use Outcomes Among Sexual and Gender Minority Individuals Living with HIV Following Residential Substance Use Treatment in Washington, DC. Alcohol Treat Q. 2023;41(4):373-385. doi: 10.1080/07347324.2023.2241419. Epub 2023 Aug 8. PMID 37886040
- [Derived] Magidson JF, Belus JM, Seitz-Brown CJ, Tralka H, Safren SA, Daughters SB. Act Healthy: A Randomized Clinical Trial Evaluating a Behavioral Activation Intervention to Address Substance Use and Medication Adherence Among Low-Income, Black/African American Individuals Living with HIV/AIDS. AIDS Behav. 2022 Jan;26(1):102-115. doi: 10.1007/s10461-021-03354-1. Epub 2021 Jun 26. PMID 34173895